CLINICAL TRIAL: NCT02570178
Title: Randomized Clinical Trial Evaluating the Effectiveness of a Primary Care Intervention Using the NintendoTM Wii Console to Improve Balance and Decrease Falls in the Elderly (EWii)
Brief Title: Effectiveness of an Intervention to Improve Balance and Decrease Falls in the Elderly (EWii)
Acronym: EWii
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PI12/01677
Record Dates: First submitted 2015-07-02; First posted 2015-10-07 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Postural Balance; Accidental Falls; Intervention Studies
Keywords: clinical trial; accidental falls; postural balance; elderly; primary Health Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- standard practice advice (No Intervention): standard practice advice
- balance training (Other): balance training using the Nintendo™ Wii console and its balance board.
  Interventions: Other: balance training

INTERVENTIONS:
Other: balance training — Participants complete 2 sessions per week for 30 minutes each, over a period of three months and are distributed in groups of four individuals carrying out the exercises at once.The groups were led by monitors who had received standardized training. Each participant was barefoot on the balance board, carrying out the different exercises in the balance area of the Wii Fit™ game, according to the indications made on the screen.Eight out of the nine balance exercises were used from the Wii Fit™ game (balance bubble, soccer heading, ski jump, table tilt, ski slalom, penguin slide, snowboard slalom, tightrope walk);.The number of repetitions of each exercise varied depending on the skill of the participants but the total time dedicated to each exercise was the same for all group participants.
  Arms: balance training

SUMMARY:
The objectives of this study are to evaluate the usefulness of an intervention utilizing the NintendoTM Wii console in order to improve balance, thereby decreasing both the fear of falling as well as the number of falls, and to evaluate the correlation between balance as determined by the console and the value obtained in the Tinetti tests and the one foot stationary test.

DETAILED DESCRIPTION:
Balance alteration is a risk factor for falls in elderly individuals that has physical, psychological and economic consequences. The objectives of this study are to evaluate the usefulness of an intervention utilizing the NintendoTM Wii console in order to improve balance, thereby decreasing both the fear of falling as well as the number of falls, and to evaluate the correlation between balance as determined by the console and the value obtained in the Tinetti tests and the one foot stationary test.

Methods/Design: This is a controlled, randomized clinical trial of individual assignment, carried out on patients over 70 years in age, from five primary care centers in the city of Mataró (Barcelona). 380 patients were necessary for the intervention group that carried out the balance board exercises in 2 sessions per week for a 3 month period, and 380 patients in the control group who carried out their usual habits. Balance was evaluated using the Tinetti test, the one foot stationary test and with the console, at the start of the study, at the end of the intervention (3 months) and one year later. Quarterly telephone follow-up was also conducted to keep track of falls and their consequences.

Discussion: The study aimed to connect the community with a technology that may be an easy and fun way to assist the elderly in improving their balance without the need to leave home or join rehabilitation groups, offering greater comfort for this population and decreasing healthcare costs since there is no need for specialized personnel.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 70 or older, of both genders,
* with the ability to walk, with or without technical assistance
* who are available for a one year period and who agree to participate in the study, signing an informed consent form

Exclusion Criteria:

* Home-bound patients
* individuals who are already receiving rehabilitation treatment on walking
* those with moderate cognitive deterioration (Pfeiffer ≥5)
* terminally ill patients
* individuals who do not have a telephone
* those with communication difficulties: cognitive and/or sensory deterioration, language barriers

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1037 (Actual)
Dates: Start 2012-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Balance calculated by the Tinetti test | change from baseline in Tinetti Test at 3 and 12 months
Balance calculated by the one footed stationary test | change from baseline in one footed stationary test at 3 and 12 months
Percentage of balance calculated by the NintendoTM Wii console | change from baseline in Percentage of balance calculated by the NintendoTM Wii console at 3 and 12 months
Fear of falling | change from baseline in FES-I at 3 and 12 months
  The Short FES-I (Falls Efficacy Scale) looks at the probability of falling in seven everyday situations. Scoring ranges from 7 to 28 points (high scores indicate a greater fear of falling)

SECONDARY OUTCOMES:
Number of falls | Change from baseline in number of falls at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Pilar Montero, MD, Principal Investigator — Catalan Health System
Locations (1):
- Jordi Gol Gurina Foundation, Barcelona, Catalonia, Spain

REFERENCES:
- [Background] Gillespie LD, Robertson MC, Gillespie WJ, Sherrington C, Gates S, Clemson LM, Lamb SE. Interventions for preventing falls in older people living in the community. Cochrane Database Syst Rev. 2012 Sep 12;2012(9):CD007146. doi: 10.1002/14651858.CD007146.pub3. PMID 22972103
- [Background] Williams MA, Soiza RL, Jenkinson AM, Stewart A. EXercising with Computers in Later Life (EXCELL) - pilot and feasibility study of the acceptability of the Nintendo(R) WiiFit in community-dwelling fallers. BMC Res Notes. 2010 Sep 13;3:238. doi: 10.1186/1756-0500-3-238. PMID 20831836
- [Background] Lister C, West JH, Cannon B, Sax T, Brodegard D. Just a fad? Gamification in health and fitness apps. JMIR Serious Games. 2014 Aug 4;2(2):e9. doi: 10.2196/games.3413. PMID 25654660
- [Derived] Montero-Alia P, Miralles-Basseda R, Lopez-Jimenez T, Munoz-Ortiz L, Jimenez-Gonzalez M, Prat-Rovira J, Albarran-Sanchez JL, Manresa-Dominguez JM, Andreu-Concha CM, Rodriguez-Perez MC, Marti-Cervantes JJ, Sanudo-Blanco L, Sanchez-Perez CA, Dolader-Olive S, Toran-Monserrat P. Controlled trial of balance training using a video game console in community-dwelling older adults. Age Ageing. 2019 Jul 1;48(4):506-512. doi: 10.1093/ageing/afz047. PMID 31081504
- [Derived] Montero-Alia P, Munoz-Ortiz L, Jimenez-Gonzalez M, Benedicto-Panell C, Altimir-Losada S, Lopez-Colomer Y, Prat-Rovira J, Amargant-Rubio JF, Jastes SM, Moreno-Buitrago A, Rodriguez-Perez MC, Teixido-Vargas C, Albarran-Sanchez JL, Candel-Gil A, Serra-Serra D, Marti-Cervantes JJ, Sanchez-Perez CA, Sanudo-Blanco L, Dolader-Olive S, Toran-Monserrat P. Study protocol of a randomized clinical trial evaluating the effectiveness of a primary care intervention using the Nintendo Wii console to improve balance and decrease falls in the elderly. BMC Geriatr. 2016 Jan 12;16:8. doi: 10.1186/s12877-015-0178-x. PMID 26796956
- See also: Percentage of balance calculated by the NintendoTM Wii console: Conducting the lame duck test which calculated how the center of gravity moves when the individual is on one foot for a maximum of thirty seconds. High percentages indicate good balance — http://www.guiasnintendo.com/2a_WII/wii_fit/wii_fit_sp/test_equilibrio.html